CLINICAL TRIAL: NCT03838991
Title: Epigenetic Regulation of Activity and Severity of Fibrous Dysplasia in Bone: mirDYS Study.
Brief Title: Epigenetic Regulation in Fibrous Dysplasia of Bone: mirDYS Study.
Acronym: MirDYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0443
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: Fibrous Dysplasia of Bone
MeSH Terms: conditions — Fibrous Dysplasia of Bone | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monostotic fibrous dysplasia (Experimental): Patients with monostotic Fibrous dysplasia.
  Interventions: Other: Blood sample; Other: Waste bone tissue
- Polyostotic fibrous dysplasia (Experimental): Patients with polyostotic Fibrous dysplasia.
  Interventions: Other: Blood sample; Other: Waste bone tissue
- Controls (Active Comparator): Control patients having a scheduled surgery for osteoarthritis.
  Interventions: Other: Blood sample; Other: Waste bone tissue

INTERVENTIONS:
Other: Blood sample — A study specific blood sample will be collected.
Other: Waste bone tissue — For 3 patients of each group, patients having a scheduled surgery, a piece of waste bone tissue will be collected after surgery.

SUMMARY:
Fibrous dysplasia of bone is a rare congenital but non-hereditary disease caused by a post-zygotic activation mutation of the GNAS gene. Patients with fibrous dysplasia may present pain and bone complications (fractures, deformities..) related to their bone lesions.

For undetermined reasons, severity and disease evolution may vary considerably from patient to patient.

Epigenetic regulation could then be involved, including micro Ribonucleic Acids (miRs).

These small non-coding micro Ribonucleic Acids are involved in the regulation of major steps of cellular processes in different pathologies, in particular in bone diseases. However, micro Ribonucleic Acids have never been studied in fibrous dysplasia.

The aim of this study is to identify micro Ribonucleic Acids significantly associated with the severity of fibrous dysplasia.

ELIGIBILITY:
Inclusion Criteria:

Control population :

* men and women,
* 18 years-old and over,
* consulting a rheumatologist or an orthopedist for arthrosis
* have scheduled surgery for hip or knee replacement surgery or any intervention involving the lower limb or upper limb.

Patients with Fibrous dysplasia:

* men and women,
* 18 years-old and over,
* with a diagnosis of fibrous dysplasia previously established by a rheumatologist.

Exclusion Criteria:

* Refusal to participate in the study
* Long- term corticosteroids treatment (> 3 months)
* Treated osteoporosis
* Chronic inflammatory rheumatism (rheumatoid arthritis, psoriasic arthritis, spondyloarthropathy)
* Collagen disease (osteogenesis imperfecta…)
* Paget's disease, benign bone tumors
* Uncontrolled hypo/hyper-thyroidism, hypo/hyper-parathryoidism
* Severe renal impairment (GFR < 30 ml/min/1.73m2)
* Cancer or bone metastases (current or in the past two years)
* Paget disease, benign bone tumor (osteoid osteoma, enchondroma …)
* Malabsorptive disease (Celiac disease, Whipple's disease, intestinal bypass, short bowel syndrome) and inflammatory bowel disease
* Pregnant women or lactating
* Psychiatric disorders
* Difficulty in understanding French
* Not a beneficiary of french social security
* Patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of micro Ribonucleic acids expression in the serum | At inclusion
  The objective is to identify specific microRibonucleic acids expressed in serum of patients using NGS (Next Generation Sequencing).
Evaluation of micro Ribonucleic acids expression in the bone tissue | At inclusion
  The objective is to identify specific micro Ribonucleic acids expressed in bone tissue obtained from surgery (patients having a scheduled surgery for osteoarthritis or fibrous dysplasia) using NGS (Next Generation Sequencing)

SECONDARY OUTCOMES:
Comparison of micro Ribonucleic acids expression | Time of realization of the analyzes, an average of 6 months
  The objective is to compare nature and level of expression of the micro Ribonucleic acids identify by NGS (Next Generation Sequencing) in bone tissue and serum between the 3 groups of subjects: monostotic Fibrous Dysplasia, polyostotic Fibrous Dysplasia and controls (controls are patients with osteoarthritis).
Validation of micro Ribonucleic acids identified by NGS (Next Generation Sequencing) in blood samples | Time of realization of the analyzes, an average of 6 months
  The objective is to validate expression of micro Ribonucleic acids identified by NGS (Next Generation Sequencing) in blood samples of patients from 4 pre-existing cohorts : a fibrous dysplasia cohort (PERIOSDYS) and 3 cohorts of control patients (OFELY and MODAM for women, STRAMBO for men).
  For that the expression of the significant micro Ribonucleic acids identified by NGS (Next Generation Sequencing) in sera of patients with monostotic and polyostotic fibrous dysplasia versus control patients will be measured by RT-qPCR (Reverse Transcription Quantitative Polymerase Chain Reaction) and then these results will be compared with same analysis on blood samples of patients from the 4 pre-existing cohorts.
Association between micro Ribonucleic acids and severity of fibrous dysplasia. | Time of realization of the analyzes, an average of 6 months
  Association between expression of significant micro Ribonucleic acids in patients with fibrous dysplasia with the severity of the disease will be studied by statistics analysis.
  Severity of fibrous dysplasia will be evaluated with clinical, biological and radiological data extracted from patients' medical records (Easily software) and from the CEMARA database (fibrous dysplasia database).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie & INSERM U1033, Pavillon F, Hopital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Legrand MA, Millet M, Merle B, Rousseau JC, Hemmendinger A, Gineyts E, Sornay-Rendu E, Szulc P, Borel O, Croset M, Chapurlat R. A Signature of Circulating miRNAs Associated With Fibrous Dysplasia of Bone: the mirDys Study. J Bone Miner Res. 2020 Oct;35(10):1881-1892. doi: 10.1002/jbmr.4111. Epub 2020 Jul 21. PMID 32526052